CLINICAL TRIAL: NCT03054116
Title: Airflow Perturbation Device (APD) for the Evaluation of Pulmonary and Sleep Disorders
Status: Completed | Type: Observational
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Aaron B. Holley, Aaron Holley, MD, Chief of Sleep Medicine, Walter Reed National Military Medical Center
Other Study IDs: 383145
Record Dates: First submitted 2017-02-08; First posted 2017-02-15 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Airway Obstruction
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Airflow pertubation device — Participants have airway resistance measured at the mouth by tidal breathing into a mouth-piece connected to the airflow perturbation device.
  Other Names: APD

SUMMARY:
In a prospective, observational study the investigators compared resistance values measured using the airway perturbation device (APD) to impulse oscillometry and spirometry. The investigators also created reference equations for normal APD resistance ranges using the data from clinically normal volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects > 18 years
* Referred for PFTs and/or PSG at WRNMMC
* All races and ethnicities will be included
* Pregnant women will be included

Exclusion Criteria:

* < 18 years of age
* If mental status is questionable, the patient will be excluded at the discretion of the consenting provider
* Unable/unwilling to follow the directions necessary for APD use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients referred to the Walter Reed NNMC pulmonary clinic mixed with clinically normal volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2014-08-31 (Actual); Study Completion 2014-08-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with APD correlation > 0.5 with spirometry | At enrollment
  Respiratory resistance ( cm H20/L/s) measured with APD correlated with volumes (in liters) measured by spirometry.

SECONDARY OUTCOMES:
Number of participants with APD correlation > 0.5 with impulse oscillometry | At enrollment
  Respiratory resistance (cm H20/L/s) measured with APD correlated with resistance (cm H20/L/s) measured using impulse oscillometry

IPD SHARING:
Plan to Share IPD: No